CLINICAL TRIAL: NCT00362908
Title: Diets for Dyslipidemia in the Metabolic Syndrome
Brief Title: Effects of Low and Moderate Fat Diets on Lipids, Inflammation and Vascular Reactivity in the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Pathmaja Paramsothy, MD, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 29854-B; R01HL083117 (NIH); 422
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Metabolic Syndrome X; Dyslipidemias
Keywords: Obesity; Hypertension; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Dyslipidemias; Obesity; Hypertension; Insulin Resistance | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Subjects consume study diets in the following order:
  1. Diet 1 (20% fat diet) for 1 month with all food provided,
  2. American Heart Association Step I Diet for 1 month at home, and
  3. Diet 2 (40% fat diet) for 1 month with all food provided and then continue to follow this diet for an additional 4 months at home.
  Interventions: Behavioral: Moderate Fat and Moderate Carbohydrate Diet; Behavioral: Low Fat and High Carbohydrate Diet
- Group 2 (Active Comparator): Subjects consume study diets in the following order:
  1. Diet 2 (40% fat diet) for 1 month with all food provided,
  2. American Heart Association Step I Diet for 1 month at home, and
  3. Diet 1 (20% fat diet) for 1 month with all food provided and then continue to follow this diet for an additional 4 months at home.
  Interventions: Behavioral: Moderate Fat and Moderate Carbohydrate Diet; Behavioral: Low Fat and High Carbohydrate Diet

INTERVENTIONS:
Behavioral: Moderate Fat and Moderate Carbohydrate Diet — 40% allowable fat diet (less than or equal to 7% saturated fat) consumed for 1 or 5 months
Behavioral: Low Fat and High Carbohydrate Diet — 20% fat diet (less than or equal to 7% saturated fat) consumed for 1 or 5 months

SUMMARY:
The metabolic syndrome consists of five concurrent conditions which increase risk of heart disease, stroke, and diabetes. Persons with the metabolic syndrome usually have high triglyceride and low HDL levels and are overweight. Low fat, high carbohydrate diets may not provide the same cholesterol-lowering benefits to obese individuals as they do to non-obese individuals. The purpose of this study is to compare the effects of a low fat, high carbohydrate diet versus a moderate fat, moderate carbohydrate diet on the heart, blood vessels, and cholesterol levels in individuals with metabolic syndrome.

DETAILED DESCRIPTION:
The Metabolic Syndrome is characterized by elevated insulin levels, excess body fat in the waist, and elevated levels of glucose and blood pressure, and dyslipidemia. Dyslipidemia in the Metabolic Syndrome is characterized by high levels of triglycerides, low levels of HDL cholesterol, and above average LDL and non-HDL cholesterol. Individuals with elevated LDL cholesterol have traditionally been advised to follow a low fat, high carbohydrate diet. However, research has shown that this diet does not adequately regulate cholesterol levels in individuals with dyslipidemia. A diet consisting of more moderate amounts of fats and carbohydrates may be more beneficial for individuals with the dyslipidemia of the metabolic syndrome. The purpose of this study is to compare the effects of a diet moderate in fat and carbohydrate versus a low fat, high carbohydrate diet on the cholesterol levels, inflammatory factors and vascular response in individuals with metabolic syndrome.

During the initial screening period, participants follow an American Heart Association (AHA) Step 1 diet and cholesterol levels are tested for eligibility under the criteria of the Metabolic Syndrome. Before being randomized, eligible participants have a frequently sampled intravenous glucose tolerance test (FSIVGTT), an abdominal CT scan to measure fat content in two locations and two brachial artery reactivity tests. The FSIVGTT provides information about whether participants are insulin sensitive or insulin resistant. The CT scan measures the fat content in the abdomen and the liver. The brachial artery reactivity tests measure blood flow through the brachial artery in the arm.

This 7-month study consists of two 1-month feeding periods, a rest month between the two feeding periods and a 4-month follow-up diet in a free-living setting. In Month 1, participants are randomly assigned to follow either a moderate fat, moderate carbohydrate diet or a low fat, high carbohydrate diet. Participants receive prepared food at study visits twice a week. Weight and vital signs are measured at each study visit, and blood is collected at baseline, and Weeks 3-1/2 and 4. A brachial artery reactivity test, using an ultrasound to measure artery size and blood flow in the arm, is performed twice in Week 4. In the Month 2 rest period, participants follow an AHA Step 1 diet at home. In Month 3, participants switch to the other diet and all study procedures and evaluations are repeated as in Month 1. During the following Months 4 through 7, participants continue following the second assigned diet, but are responsible for preparing their own food. They meet with a dietician once a week for 1 month to learn how to prepare meals at home. During this 4-month period, blood collection, vital sign measurements, and review of medical history and diet continue at monthly visits. At the end of Month 7, participants again undergo two brachial artery reactivity tests.

As of October, 2010, 148 were screened with 71 eligible to be randomized. Seven discontinued prior to completion and 64 completed the 7 month study. The intervention is complete and analyses are ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic Syndrome: individuals must have at least three of the following five criteria:

  1. Abdominal obesity greater than 90 cm in Asian men, greater than 102 cm in all other men, greater than 80 cm in Asian women, and greater than 88 cm in all other women
  2. Triglycerides greater than or equal to 150 mg/dL at two screening visits (Required for the purposes of this study, which focuses on the dyslipidemic phenotype)
  3. HDL cholesterol levels less than 40 mg/dL in men and less than 50 mg/dL in women
  4. Blood pressure levels greater than 130/85 mmHg or taking an allowed blood pressure medication at Visit 1 (see definition in exclusions below)
  5. Fasting glucose greater than or equal to 100mg/dL at Visit 1

Exclusion Criteria:

* LDL greater than or equal to 190 mg/dL
* Triglycerides greater than 500mg/dL at Visit 1
* Blood pressure over a mean of 150/95 at the two first visits
* Body mass index greater than 40 kg/m²
* Currently taking any lipid lowering medication other than statins
* Currently taking high doses of thiazide diuretics (greater than 50mg/day), or any other blood pressure medication in the past 4 weeks
* Use of plant sterols from sources such as Benecol or Take Control margarines in the past 4 weeks
* Use of any fish oil supplements in the week prior to screening
* Blood glucose greater than 140 mg/dL or use of diabetes medications
* Hospitalization for coronary disease in the last 6 months
* Use of nitroglycerin or other nitrates
* Unstable liver, renal, gastrointestinal or pulmonary disease or mental disease, or medically unstable for other reasons
* Alcohol intake greater than 2 drinks/day, any illegal drug use, smoking, chronic NSAID use or NSAID use within 5 days before the BAR study
* Pregnancy intended within one year or one year prior or currently lactating
* In reproductive age women, an irregular menstrual cycle (must have consistent menstrual cycle between 24 to 32 days)
* Use or expectation of use of oral or patch contraceptive
* Unable or unlikely to be able to comply with study requirements

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Non-HDL cholesterol | Measured at screening, baseline, at the beginning and end of the 1st and 2nd diet periods, and at the end of each month for four months during the diet extension
C-reactive protein | Measured at the beginning and end of the 1st and 2nd diet periods and at the end of the four month diet extension
Brachial artery reactivity | Two measurements are done at the beginning and end the 1st and 2nd diet periods and at the end of the four month diet extension

CONTACTS AND LOCATIONS:
Overall Officials: Pathmaja Paramsothy, MD, Principal Investigator — University of Washington
Locations (1):
- Northwest Lipid Research Clinic, Seattle, Washington, United States

REFERENCES:
- [Background] Knopp RH, Fish B, Dowdy A, Retzlaff B, Walden C, Rusanu I, Paramsothy P. A moderate-fat diet for combined hyperlipidemia and metabolic syndrome. Curr Atheroscler Rep. 2006 Nov;8(6):492-500. doi: 10.1007/s11883-006-0025-9. PMID 17045076
- [Result] Paramsothy P, Krieger E, Chan E, Fish B, Dowdy A, Knopp RH. Abstract 1017: Moderate vs Low Fat Diet Effects on Lipids and Inflammation in Metabolic Syndrome. Circulation, Nov 2009; 120: S426. Presented as oral abstract at AHA Annual Scientific Session November, 2009.
- [Result] Paramsothy P, Kreiger E, Chan E, Preus E, Rusanu I, Prager S, Knopp RH. Effects Of Low Fat Vs. Moderate Fat Diet On Insulin Resistance And Endothelial Function In Metabolic Syndrome. J. Am. Coll. Cardiol., March 9, 2010; 55: A58.E555. Presented as poster at ACC, Atlanta, GA. 3/10.